CLINICAL TRIAL: NCT04720196
Title: Analgesic Effect of Repetitive Transcranial Magnetic Stimulation in Painful Vasculitic Neuropathy
Brief Title: Analgesic Effect of rTMS in Vasculitic Neuropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JagiellonianU63
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Vasculitic Neuropathy
Keywords: vasculitis; neuropathy; pain; transcranial magnetic stimulation; analgesic effect
MeSH Terms: conditions — Vasculitis; Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to active and then sham stimulation or to sham and then active stimulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham stimulation will be provided by holding the stimulating coil perpendicularly to the scalp, which assures similar impression as during active stimulation but prevents significant magnetic field to reach the brain tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active repetitive transcranial magnetic stimulation (Experimental): 10 hertz (Hz) rTMS will be administered over the primary motor area. Therapy will include 5 daily sessions (on consecutive week days). In every sessions 1500 magnetic pulses of 90% of the resting motor threshold intensity will be elicited.
  Interventions: Device: Active repetitive transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation (Sham Comparator): Sham stimulation will mimic the active one except that the stimulating coil will be held perpendicularly to the scalp, which assures similar impression as the active stimulation but prevents that significant magnetic field will reach brain tissue.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation — High frequency rTMS over the primary motor area to induce the long term potentiation of primary motor areas for the muscles of upper extremity.
  Arms: Active repetitive transcranial magnetic stimulation
Device: Sham repetitive transcranial magnetic stimulation — Sham stimulation to mimic the high frequency rTMS over the primary motor area.
  Arms: Sham repetitive transcranial magnetic stimulation

SUMMARY:
Vasculitic neuropathy (VN) results from inflammation and destruction of the walls of predominantly small vessels with subsequent ischemic damage of peripheral nerves. VN is painful in vast majority of patients and the pain is intractable with pharmacotherapy in about 40% of cases. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity and is regarded as one of alternative methods to alleviate pain associated with various kind of neuropathies. The purpose of this study is to compare the effectiveness of analgesic effect of rTMS in vasculitic neuropathy with sham stimulation.

DETAILED DESCRIPTION:
Vasculitic neuropathies (VN) are a group of disorders resulting from inflammation of predominantly small vessels with destruction of their walls and subsequent ischemic damage of peripheral nerves. Neural damage may or may not coexist with the damage of other organs. Examples of conditions associated with VN include diabetes, microscopic polyangiitis, eosinophilic granulomatosis with polyangiitis (Churg-Strauss), granulomatosis with polyangiitis (Wegener's), rheumatoid arthritis, systemic lupus erythematosus and others. VN is painful in about 80% of patients of whom 40% suffer from the pain intractable with pharmacological therapy. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive method of modulation of brain plasticity. In this method, series of magnetic stimuli are delivered to the cerebral cortex, where they turn to electric current and depolarize repetitively the targeted neurons. If the stimulation is repeated during subsequent days it is capable to modify the activity of targeted cortical area for weeks or even months and by this way to achieve therapeutic effect. rTMS is widely regarded as one of alternative methods to alleviate pain associated with various kind of neuropathies. The purpose of this study is to compare the effectiveness of analgesic effect of rTMS in vasculitic neuropathy with sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vasculitic neuropathy
* Neuropathic pain of constant severity since not less than a month and requiring use of analgesics more than once a week
* Score of 30 milimeter or more on the 100 milimeter visual analog scale of pain intensity at inclusion

Exclusion Criteria:

* Severe depression
* Personality disorders and other psychiatric conditions, which could disturb the participation in the study
* Cognitive deficits, which could disturb the participation in the study
* Contraindications for rTMS as listed by the Guidelines of the International Federation of Clinical Neurophysiology (Rossi et al. 2009) i.e. seizure in the past, epilepsy, presence of magnetic material in the reach of magnetic field, pregnancy, likelihood to get pregnant, intracranial electrodes, cardiac pacemaker or intracardiac lines, frequent syncopes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Severity Scale after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Total score 10, with higher scores representing more severe pain. Change from baseline score in the Numeric Pain Severity Scale to the measurement taken after finishing rTMS.
Numeric Pain Severity Scale First Follow Up | Before rTMS, two weeks after finishing rTMS
  Total score 10, with higher scores representing more severe pain. Change from baseline score in the Numeric Pain Severity Scale to the measurement taken two weeks after finishing rTMS.
Numeric Pain Severity Scale Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Total score 10, with higher scores representing more severe pain. Change from baseline score in the Numeric Pain Severity Scale to the measurement taken four weeks after finishing rTMS.
Visual Analog Scale of Pain Severity | Through study completion, an average of 10 weeks
  An analog scale of the length of 100 milimeter. Total score of 100, with higher scores representing more severe pain. Change through the study.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Total score 64, with higher scores representing more severe depression. Change from baseline score in the Hospital Anxiety and Depression Scale to the measurement taken after finishing rTMS.
Hospital Anxiety and Depression Scale First Follow Up | Before rTMS, two weeks after finishing rTMS
  Total score 64, with higher scores representing more severe depression. Change from baseline score in the Hospital Anxiety and Depression Scale to the measurement taken two weeks after finishing rTMS.
Hospital Anxiety and Depression Scale Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Total score 64, with higher scores representing more severe depression. Change from baseline score in the Hospital Anxiety and Depression Scale to the measurement taken four weeks after finishing rTMS.
36-Item Short Form Health Survey after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Total score, range 0 to 800, with lower values representing a worse outcome. Change from baseline score in the 36-Item Short Form Health Survey to the measurement taken after finishing rTMS.
36-Item Short Form Health Survey First Follow Up | Before rTMS, two weeks after finishing rTMS
  Total score, range 0 to 800, with lower values representing a worse outcome. Change from baseline score in the 36-Item Short Form Health Survey to the measurement taken two weeks after finishing rTMS.
36-Item Short Form Health Survey Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Total score, range 0 to 800, with lower values representing a worse outcome. Change from baseline score in the 36-Item Short Form Health Survey to the measurement taken four weeks after finishing rTMS.
Quality of Life in Neurological Disorders (Neuro-QoL) Upper Extremity Function after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Total score, range 0 to 100, with lower values representing a worse outcome. Change from baseline score in Neuro-Qol Upper Extremity Function to the measurement taken after finishing rTMS.
Quality of Life in Neurological Disorders (Neuro-QoL) Upper Extremity Function First Follow Up | Before rTMS, two weeks after finishing rTMS
  Total score, range 0 to 100, with lower values representing a worse outcome. Change from baseline score in Neuro-Qol Upper Extremity Function to the measurement taken two weeks after finishing rTMS.
Quality of Life in Neurological Disorders (Neuro-QoL) Upper Extremity Function Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Total score, range 0 to 100, with lower values representing a worse outcome. Change from baseline score in Neuro-Qol Upper Extremity Function to the measurement taken four weeks after finishing rTMS.
Assessment of pain threshold to electric stimuli after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Electrocutaneus stimulation with gradually increasing intensity from 0mA until a patient reports that the sensation has become painful. Change from baseline pain threshold to the measurement taken after finishing rTMS.
Assessment of sensory threshold to electric stimuli after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Electrocutaneus stimulation with gradually increasing intensity from 0mA until a patient reports the first nonpainful tactile sensation. Change from baseline sensory threshold to the measurement taken after finishing rTMS.
Assessment of pain threshold to electric stimuli First Follow Up | Before rTMS, two weeks after finishing rTMS
  Electrocutaneus stimulation with gradually increasing intensity from 0mA until a patient reports that the sensation has become painful. Change from baseline pain threshold to the measurement taken two weeks after finishing rTMS.
Assessment of sensory threshold to electric stimuli First Follow Up | Before rTMS, two weeks after finishing rTMS
  Electrocutaneus stimulation with gradually increasing intensity from 0mA until a patient reports the first nonpainful tactile sensation. Change from baseline sensory threshold to the measurement taken two weeks after finishing rTMS.
Assessment of pain threshold to electric stimuli Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Electrocutaneus stimulation with gradually increasing intensity from 0mA until a patient reports that the sensation has become painful. Change from baseline pain threshold to the measurement taken four weeks after finishing rTMS.
Assessment of sensory threshold to electric stimuli Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Electrocutaneus stimulation with gradually increasing intensity from 0mA until a patient reports the first nonpainful tactile sensation. Change from baseline sensory threshold to the measurement taken four weeks after finishing rTMS.
Assessment of cold sensation threshold to cold stimuli after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Stimulation with cold temperature stimuli, gradually colder, starting from from 32 degree Celcius until patient will report that he feels cold. Change from baseline cold sensation threshold to the measurement taken after finishing rTMS.
Assessment of pain threshold to cold temeprature stimuli after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Stimulation with cold temperature stimuli, gradually colder, starting from 32 degree Celcius until patient starts to perceive stimuli as painful. Change from baseline pain threshold to the measurement taken after finishing rTMS.
Assessment of cold sensation threshold to cold temeprature stimuli First Follow Up | Before rTMS, two weeks after finishing rTMS
  Stimulation with cold temperature stimuli, gradually colder, starting from from 32 degree Celcius until patient will report that he feels cold. Change from baseline cold sensation threshold to the measurement taken two weeks after finishing rTMS.
Assessment of pain threshold to cold temeprature stimuli First Follow Up | Before rTMS, two weeks after finishing rTMS
  Stimulation with cold temperature stimuli, gradually colder, starting from 32 degree Celcius until patient starts to perceive stimuli as painful. Change from baseline pain threshold to the measurement taken two weeks after finishing rTMS.
Assessment of cold sensation threshold to cold temeprature stimuli Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Stimulation with cold temperature stimuli, gradually colder, starting from from 32 degree Celcius until patient will report that he feels cold. Change from baseline cold sensation threshold to the measurement taken four weeks after finishing rTMS.
Assessment of pain threshold to cold temeprature stimuli Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Stimulation with cold temperature stimuli, gradually colder, starting from 32 degree Celcius until patient starts to perceive stimuli as painful. Change from baseline pain threshold to the measurement taken four weeks after finishing rTMS.
Assessment of warmth sensation threshold to warm temeprature stimuli after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Stimulation with warm temperature stimuli, gradually warmer, starting from from 32 degree Celcius until patient will report that he feels warmth. Change from baseline warmth sensation threshold to the measurement taken after finishing rTMS.
Assessment of pain threshold to warm temeprature stimuli after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Stimulation with warm temperature stimuli, gradually warmer, starting from 32 degree Celcius until patient starts to perceive stimuli as painful. Change from baseline pain threshold to the measurement taken after finishing rTMS.
Assessment of warmth sensation threshold to warm temeprature stimuli First Follow Up | Before rTMS, two weeks after finishing rTMS
  Stimulation with warm temperature stimuli, gradually warmer, starting from from 32 degree Celcius until patient will report that he feels warmth. Change from baseline warmth sensation threshold to the measurement taken two weeks after finishing rTMS.
Assessment of pain threshold to warm temeprature stimuli First Follow Up | Before rTMS, two weeks after finishing rTMS
  Stimulation with warm temperature stimuli, gradually warmer, starting from 32 degree Celcius until patient starts to perceive stimuli as painful. Change from baseline pain threshold to the measurement taken two weeks after finishing rTMS.
Assessment of warmth sensation threshold to warm temeprature stimuli Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Stimulation with warm temperature stimuli, gradually warmer, starting from from 32 degree Celcius until patient will report that he feels warmth. Change from baseline warmth sensation threshold to the measurement taken four weeks after finishing rTMS.
Assessment of pain threshold to warm temeprature stimuli Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Stimulation with warm temperature stimuli, gradually warmer, starting from 32 degree Celcius until patient starts to perceive stimuli as painful. Change from baseline pain threshold to the measurement taken four weeks after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the index finger flexion after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Change from baseline strength of the index finger flexion to the measurement taken after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the foot extension after rTMS | Before rTMS, immediately after (on same day) finishing rTMS.
  Change from baseline strength of the foot extension to the measurement taken after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the index finger flexion First Follow Up | Before rTMS, two weeks after finishing rTMS
  Change from baseline strength of the index finger flexion to the measurement taken two weeks after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the foot extension flexion First Follow Up | Before rTMS, two weeks after finishing rTMS
  Change from baseline strength of the foot extension to the measurement taken two weeks after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the index finger flexion Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Change from baseline strength of the index finger flexion to the measurement taken four weeks after finishing rTMS.
Bilateral Dynamometric Assessment of the strength of the foot extension Second Follow Up | Before rTMS, four weeks after finishing rTMS
  Change from baseline strength of the index foot extension to the measurement taken four weeks after finishing rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Brączyk, MS, Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Neurology, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Yes
After completing the study, the age and gender of participants as well as the scores and results of all outcome measurements made at baseline, after rTMS, at the first and at the second follow up will be made available to other researchers on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the study results will be published.
Access Criteria: On request send by e-mail: jakub.antczak@uj.edu.pl

REFERENCES:
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552